CLINICAL TRIAL: NCT05217563
Title: Reframing Needle-Related Pain: Randomized Clinical Trial of a Parent-Led Memory-Reframing Intervention
Brief Title: Reframing Needle-related Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: University of Calgary (Other)
Collaborators: Alberta Children's Hospital Research Institute (Other); Solutions for Kids in Pain (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB21-1997
Record Dates: First submitted 2021-12-14; First posted 2022-02-01 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-02

CONDITIONS: Pain, Procedural
Keywords: pediatric pain; parents; needle-related pain; vaccination injection; memory for pain; memory-reframing intervention
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Parallel arm design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care (No Intervention): Standard Care Control Group (Group 1). Parents in the standard care control group will receive a pamphlet containing evidence-based information on needle pain management. Parents in the standard care control group will not receive any information regarding pain memory reframing, nor will they be encouraged to talk about their children's pain vaccine injection experience. Parents in the standard care control group will receive text/email reminders to use needle pain management strategies before each second vaccination appointment.
- Intervention Group (Pamphlet and video only) (Active Comparator): Intervention Group (Group 2; Pamphlet and video Only). Parents in this intervention group will receive a pamphlet containing evidence-based information on needle pain management and a pamphlet summarizing memory reframing principles. The pamphlet will have a link to a video summarizing the memory reframing strategies.
  Interventions: Behavioral: Memory-reframing intervention (Reframe the Pain)
- Intervention Group (Pamphlet, video, and verbal Instructions). (Active Comparator): Intervention Group (Group 3; Handout and Verbal Instructions). Parents in this intervention group will receive a pamphlet containing evidence-based information on needle pain management, a pamphlet summarizing memory reframing principles (with a video link), and verbal instructions on how to use the intervention principles with their children. The instructions will be provided via telephone or video conferencing and will last approximately 10 to 15 minutes. Trained graduate students or post-doctoral fellows will deliver the instructions. Similar to previous interventions, to boost mastery of the material, the researcher will provide suggestions for specific questions and remarks to make while reminiscing. The instructions will be audio-recorded to allow fidelity coding.
  Interventions: Behavioral: Memory-reframing intervention (Reframe the Pain)

INTERVENTIONS:
Behavioral: Memory-reframing intervention (Reframe the Pain) — Parents will be taught to reminisce with their children about the vaccination experience by emphasizing positive aspects of the child's pain memory, using less utterances about pain and fear, correcting negative exaggerations in memory, and enhancing children's self-efficacy regarding their ability to cope with pain (e.g., when children used coping methods such as deep breathing, highlighting that they were brave). Parents will be instructed to reminisce with their children about the vaccine experience using the intervention strategies. Parents in the intervention groups will receive text/email reminders to use needle pain management strategies before each second vaccination appointment. Additionally, parents randomized to the intervention groups will receive text/email reminders approximately once every two weeks to use the memory-reframing principles until the second vaccination appointment.
  Arms: Intervention Group (Pamphlet and video only); Intervention Group (Pamphlet, video, and verbal Instructions).

SUMMARY:
The present research study aims to examine the efficacy of a brief parent-led memory reframing intervention to foster more adaptive (i.e., more accurate and positive) pain memories and less future needle pain and fear for a two-series needle procedure (approved vaccines to protect against COVID-19; e.g., BioNTech Pfizer). The intervention will draw from recent data and extant memory reframing and narrative-based intervention techniques to promote more accurate/positive pain memories by teaching parents more adaptive styles of reminiscing with their children about a needle procedure (i.e., a COVID-19 vaccine).

DETAILED DESCRIPTION:
Pain is a common experience in childhood. Healthy children who adhere to recommended medical care undergo up to 20 painful procedures by the age of 5. Pain from, and fear of, medical experiences are neither short lasting or benign and can influence children long after the painful stimulus is removed. Children's memories of needle-related, experimental, post-surgical, and procedural pain are a powerful predictor of future pain experiences, and are sometimes more influential to future pain than the initial experience of pain itself. Memory is susceptible to distortion. Negative biases in pain memories (i.e., recalling higher levels of pain as compared to initial pain report) are associated with higher subsequent pain, distress, and worse medical compliance. Children who are more anxious and who experience greater pain are more likely to develop negatively biased pain memories, which then leads to greater fear and pain at subsequent pain experiences. Parents and adolescents who think in more catastrophic ways about child pain tend to develop more negatively biased pain memories months later. In particular, adolescents who felt helpless in the face of pain (lack of self-efficacy in their ability to deal with pain) prior to surgery went on to develop more negatively-biased memories. Moreover, parents' catastrophic thinking about child pain was found to be the single most important predictor of children's memory biases and subsequent pain trajectories. It has been suggested that parental and child anxiety lead to memory biases because of the ways in which parents and children talk about pain following painful events (e.g., by emphasizing threatening aspects of the experience). Needle fear and vaccine hesitancy have also been argued to play an important role in children's and parent reactions to needle pain.

There have only been a few studies examining memory reframing interventions in the context of children's recall of (needle) pain. In a systematic review, existing trials of memory reframing interventions were found to be efficacious in reducing negative memory biases, which is thought to be due to increases in self-efficacy. Indeed, parent-child language-based interactions about past negative events play a powerful role in how autobiographical memories of those events are subsequently retrieved and reframed. Parent-child narrative style also influences children's coping and psychological functioning. Young children whose parents are topic-extending and elaborative (e.g., who ask open-ended questions to pull for richer, more detailed accounts of the past) and who use emotional language, have children who are more accurate and detailed in recalling their pasts, which is adaptive.

Recent data provides compelling evidence that parents who reminisce with their children about surgery using a particular style (e.g., more elaborative, less topic-switching) and content (e.g., less content about pain, fear, medical procedures; more explanations) have children who later remember post-surgical pain in a more accurate and positively biased way. In a recently published pilot randomized controlled trial, the investigators demonstrated that a parent-led memory-reframing intervention is efficacious in reducing negative biases in children's memories for post-surgical pain. However, the intervention has not been examined in the context of needle procedures. The potential impact of the intervention on children's future pain experiences has not yet been examined. Finally, the parent-led memory-reframing intervention has only been tested in children aged 4 to 7 years. A recent RCT has demonstrated that a parent-led memory-reframing intervention is feasible and acceptable in youth aged 10 to 18 years undergoing major surgeries. Yet, the intervention efficacy for needle pain in older children is unknown.

The present research study aims to examine the efficacy of a brief parent-led memory reframing intervention to foster more adaptive (i.e., more accurate and positive) pain memories and less future needle pain and fear for a two-series needle procedure (approved vaccines to protect against COVID-19; e.g., BioNTech Pfizer). The intervention will draw from the recent data and extant memory reframing and narrative-based intervention techniques to promote more accurate/positive pain memories by teaching parents more adaptive styles of reminiscing with their children about a needle procedure (i.e., a COVID-19 vaccine). All participating parents will receive evidence-based information on pain management techniques. Parents randomized to the control group will receive a pamphlet outlining pain management strategies. Parents randomized to the intervention group will receive this same pamphlet and additionally receive a pamphlet and video link with memory-reframing instructions based on a previously published study. The third group will receive the pamphlet outlining pain management strategies, the memory-reframing pamphlet and video, as well as brief verbal instructions via telephone or zoom on how to deliver the intervention to their children. Parents randomized to the intervention groups will receive text reminders to use the intervention after the vaccine injection.

This study will be the first to test a brief, parent-led intervention aimed at changing the way children recall their pain after a needle procedure and examine the impact of the intervention on children's future needle pain intensity and fear at a second vaccine injection. This study has great potential to contribute an accessible and feasible pediatric pain management intervention and foster more adaptive pain trajectories and medical experiences in childhood.

Novelty and urgency. At this moment in time, a global health crisis is unfolding. The need for vaccinating all population, including children, must outpace the spread of COVID-19 and its variants. On November 19, 2021, Health Canada approved the Pfizer vaccine for use in children aged 5 to 11 years in Canada. Only days later parents began booking their children for these vaccinations. These vaccinations have already started. There is a considerable challenge that needs to be overcome. Two thirds of children report having needle fears. In the wake of misinformation and concerns around needle fears and needle pain, vaccine hesitancy is growing. Approximately 7-8% of parents delay or avoid having their child vaccinated due to their child's fear of needles. One way to conquer the fears increase vaccine confidence is by providing children and parents with simple yet effective strategies for managing needle pain and fear and fostering more positive memories of these procedures to improve the rate of subsequent vaccine injections. This project aims to achieve these goals. The need to do this work is urgent.

STUDY AIMS

This 3-arm randomized controlled trial seeks to achieve the following:

Primary Aims

1. To examine the efficacy of a parent-led memory reframing intervention on children's memories for pain associated with vaccine needle injections.

   Hypothesis 1. The magnitude of the intervention effect will differ depending on the group allocation. Children in the intervention group that will receive the pain management and memory intervention pamphlets (with a video link) and verbal instructions (Group 3) will recall needle-related pain in a more accurate or positively biased way as compared to the intervention group that will receive the pain management and memory intervention pamphlets (with a video link) (Group 2), followed by the pain management pamphlet only (Group 1).
2. To examine the efficacy of a parent-led memory reframing intervention on reducing children's future pain intensity and pain-related fear associated with vaccine needle injections.

   Hypothesis 2. The magnitude of the intervention effect will differ depending on the group allocation. Children in the intervention group that will receive the pain management and memory intervention pamphlets (with a video link) and verbal instructions (Group 3) will report lower levels of pain intensity and pain-related fear associated with the second vaccine injection shot as compared to the intervention group that will receive the pain management and memory pamphlets (with a video link) only (Group 2), followed by the pain management pamphlet only (Group 1).

   Secondary Aims
3. To examine the acceptability, feasibility, and adherence of different modes of intervention delivery.

   Hypothesis 3. There will be no significant differences in acceptability and feasibility across the two pamphlet(s) (with a video link) only intervention groups (Groups 2 and 3). Group 2 (pain management and memory intervention pamphlets (with a video link) only) would be lower in adherence, as compared to Group 3 (pain management and memory pamphlets + verbal instructions).
4. To examine the changes in children's and parent self-efficacy and children's expected levels of pain and pain-related fear.

Hypothesis 4. The magnitude of the intervention effect will differ depending on the group allocation. Children in the intervention group that will receive the pain management and memory intervention pamphlets (with a video link) and verbal instructions (Group 3) will report higher levels of self-efficacy and lower levels of expected pain and pain-related fear (prior to the second vaccination injection), as compared to children in the that receive the pain management and memory intervention pamphlets (with a video link) only (Group 2), followed by the pain management pamphlet only (Group 1). Similarly, parents in the intervention group that will receive the pain management and memory intervention pamphlets and verbal instructions (Group 3) will report higher levels of self-efficacy as compared to children in the intervention group that will receive the pain management and memory pamphlets (with a video link) only (Group 2), followed by the pain management pamphlet only (Group 1).

Procedure

Participants will be recruited via advertising the study on social media (e.g., Facebook, Twitter) and through KT collaborators (e.g., Solutions for Kids in Pain [SKIP]). Families interested in participating in the study will contact the research team and be screened for eligibility via telephone by the research staff. Eligible participants will provide verbal consent and will be sent a written consent form via a secure online software (i.e., REDCap) several days prior to the first vaccine appointment. Caregivers will provide consent for the child's participation; children, who are 7 years old or over or turn 7 during participation in the study, will provide assent. Participants will also complete baseline questionnaires assessing past child's experiences with needle procedures, child's and parent trait anxiety, needle fears, parent catastrophizing about child's pain, and vaccine hesitancy. Caregivers will report socio-demographic information.

Upon completion of the consent form, parents will be randomized into one of three groups using a random numbers generator. Parents in all three groups will receive a pamphlet with evidence-based information regarding needle pain management (Pain Management Pamphlet). Caregivers randomized to the two memory intervention groups (Groups 2 & 3) will also receive the latter pain management pamphlet and a pamphlet outlining the memory reframing principles and strategies (Memory Reframing Pamphlet with a video link; the video summarizes the memory reframing principles and is available at https://www.youtube.com/watch?v=lvCabG6_ekI&ab_channel=MegFoundationforPain). Caregivers randomized to the intervention group with additional instructions from a researcher (Group 3) will receive a telephone or video conference call in addition to the intervention pamphlet. During the call, a trained researcher (i.e., a graduate student or a post-doctoral fellow) will provide brief 10- to 15-minute verbal instructions on how to use memory-reframing principles with their child (Intervention Script). Randomization will be conducted by an external researcher using a computer random number generator.

On the day of the first vaccine appointment, caregivers will receive an online survey link to have children report their pain intensity and pain-related fear ratings after the vaccine injection using validated measures (described below). All parents will receive reminders to use evidence-based needle pain management prior the vaccine appointments. Parents randomized to the intervention groups will receive a text or an email reminder to use the memory-reframing strategies after the first vaccine injection. Reminders to use memory-reframing strategies will be sent once every two weeks until the second vaccine appointment.

Seven to ten days after the first vaccine injection, children will complete an established memory interview5 via telephone or video conference with a researcher blinded to group allocation. During the interview, children will report their memories for pain intensity and pain-related fear using the same measures as before, however this time based on recall. Children will also report how much pain intensity and pain-related fear they expect that they will experience during the second vaccine injection.

On the day of the second vaccine appointment, caregivers will receive an online survey link to have children report their pain and pain-related fear ratings after the vaccine injection using the same validated measures as before. Parents will report what pain management and memory reframing techniques they have used.

Following study completion, parents randomized to the intervention groups will complete brief measures of intervention acceptability. Forty parents randomized to the memory intervention groups (20 in each group) will be invited to participate in a brief semi-structured interview to provide their feedback on intervention. Parents in the control group will receive a pamphlet and video with memory-reframing principles after they complete the study.

ELIGIBILITY:
Inclusion Criteria: A child will be eligible to participate if they

* are aged between 4 and 11 years old at the time of the recruitment;
* plan to receive a two-dose COVID-19 vaccine;
* are able to understand and speak English;
* have at least one of their caregivers' consent to participate in the study, and this caregiver is able to speak and read English
* have Internet access.

Exclusion Criteria:

* serious developmental disabilities (e.g., Autism Spectrum Disorder) or speech/language delays, as it may make it difficult for the participants to complete all necessary study tasks (e.g., assent, memory interview);
* child's or caregiver's inability to speak and/or understand English

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Memory for pain during the first vaccination | 7 to 10 days after the first vaccination appointment
  Children will be asked to recall the first vaccination appointment and complete a pain intensity rating scale (i.e., Faces Pain Scale-Revised; range of scores 0 to 10; higher scores mean higher levels of pain) based on their memories of that time period. Biases in memory will be defined as the deviation in recalled and initial/experienced pain reports. Similar to our previous research, statistical models predicting pain memories will control for initial pain ratings that correspond to each memory question. Negatively-biased pain memories will be defined as children who remember more pain as compared to their initial pain reports. Positively biased pain memories will be defined as recalled pain that is less than initial pain reports. Accurate memories reflect no difference between recalled and experienced levels of pain.
Memory for pain-related fear during the first vaccination | 7 to 10 days after the first vaccination appointment
  Children will be asked to recall the first vaccination appointment and complete a pain-related fear rating scale (i.e., Children's Fear Scale; CFS; range of scores 0 to 4; higher scores mean higher levels of pain-related fear) based on their memories of that time period. Biases in memory will be defined as the deviation in recalled and initial/experienced pain-related fear reports. Similar to our previous research, statistical models predicting pain-related fear memories will control for initial pain-related fear ratings that correspond to each memory question. Negatively-biased memories will be defined as children who remember more pain-related fear as compared to their initial pain-related fear reports. Positively biased pain-related fear memories will be defined as recalled pain-related fear that is less than initial pain-related fear reports. Accurate memories reflect no difference between recalled and experienced levels of pain-related fear.
Child pain during the second vaccination | 6 to 8 weeks after the first vaccination appointment (subject to change depending on the Canada Health guidelines)
  Pain intensity will be assessed using a well-validated single-item faces pain scale (Faces Pain Scale-Revised; FPSR; range of scores 0 to 10; higher scores mean higher levels of pain) by children
Child pain-related fear during the second vaccination | 6 to 8 weeks after the first vaccination appointment (subject to change depending on the Canada Health guidelines)
  Children's pain-related fear will be assessed using the Children's Fear Scale (CFS; range of scores 0 to 4; higher scores mean higher levels of pain-related fear).

SECONDARY OUTCOMES:
Child self-efficacy | Baseline and 7 to 10 days after the first vaccination appointment
  Children will rate their pain-related self-efficacy. Children will use a 11-point NRS to assess "How well do you think you will do when you get your second COVID vaccine shot?". The scale will range from "0 = not well at all" to "10 = very well". Higher scores mean higher levels of pain-related self-efficacy.
Child and parent self-efficacy | Baseline and 7 to 10 days after the first vaccination appointment
  Parents will rate their pain-related self-efficacy. Parents will rate their self-efficacy by answering "How well do you think you will be able to help your child at their second COVID vaccine shot?" on a 0-10 Numerical Rating Scale ranging from "0 = not well at all" to "10 = very well". Higher scores mean higher levels of pain-related self-efficacy.
Feasibility of intervention (i.e., how many participants assigned to intervention groups received the intervention) | Baseline, pre-intervention, post-intervention, follow-up (i.e., 6 to 8 weeks after the first vaccination appointment)
  Feasibility will be assessed using study recruitment/enrollment statistics, completion of the study elements; and researchers' and parents' ratings of parents' motivation to learn, understanding of the intervention, and parent-researcher rapport (for group receiving verbal instructions only) rated on 11-point Likert scales. The range of scores is 0 to 10; higher scores mean higher feasibility.
Acceptability (i.e., participants' perception of the intervention applicability and usefulness, as well as their satisfaction with the intervention) | 6 to 8 weeks after the first vaccination appointment (subject to change depending on the Canada Health guidelines)
  Acceptability will be assessed at study completion (i.e., after memory interviews). The parent-report 9-item Treatment Evaluation Inventory-Short Form (TEI-SF) will be used to assess parental acceptability and satisfaction with the intervention. The scores range from 9 to 45; higher scores mean higher levels of treatment acceptability.
Adherence | 6 to 8 weeks after the first vaccination appointment (subject to change depending on the Canada Health guidelines)
  After the second vaccination appointment, parents will self-report their use of different pain management and memory-reframing techniques.
Expected pain | 7 to 10 days after the first vaccination appointment
  Children will rate how much pain they expect to experience during their second vaccine injection using the pain scale described above (i.e., FPS-R; range of scores 0 to 10; higher scores mean higher levels of pain)
Expected pain-related fear | 7 to 10 days after the first vaccination appointment
  Children will rate how much pain-related fear they expect to experience during their second vaccine injection using the fear scale described above (i.e., CFS; range of scores 0 to 4; higher scores mean higher levels of pain-related fear).

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Noel, PhD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided